CLINICAL TRIAL: NCT06363552
Title: A Study to Evaluate the Preliminary Safety and Efficacy of SC0191 as Single Agent or in Combination With Bevacizumab or 5-FU/LV in Advanced Colorectal Cancer
Brief Title: A Study of SC-0191 in Subjects With Metastatic Colorectal Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianshu Liu (Other)
Responsible Party: Sponsor-Investigator, Tianshu Liu, Director of Oncology Department, Shanghai Zhongshan Hospital
Organization: Shanghai Zhongshan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WETARI
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SC0191 (Experimental)
  Interventions: Drug: SC0191
- SC0191 + Bevacizumab (Experimental)
  Interventions: Drug: SC0191 + Bevacizumab
- SC0191 + 5-FU/LV (Experimental)
  Interventions: Drug: SC0191 + 5-FU/LV

INTERVENTIONS:
Drug: SC0191 — The SC0191 tablet is taken orally at a dose of 300mg once daily. Each treatment cycle consists of 28 days. Medication is administered on days 1 to 3, days 8 to 10, days 15 to 17, and days 22 to 24 of each cycle.
  Arms: SC0191
Drug: SC0191 + Bevacizumab — 1. The SC0191 tablet is taken orally at a dose of 300mg once daily. Each treatment cycle consists of 28 days. Medication is administered on days 1 to 3, days 8 to 10, days 15 to 17, and days 22 to 24 of each cycle.
  2. Bevacizumab injection is administered intravenously at a dose of 5mg/kg on day 1 and day 15 of each treatment cycle.
  Arms: SC0191 + Bevacizumab
Drug: SC0191 + 5-FU/LV — 1. The SC0191 tablet is taken orally at a dose of 300mg once daily. Each treatment cycle consists of 28 days. Medication is administered on days 1 to 3, days 8 to 10, days 15 to 17, and days 22 to 24 of each cycle.
  2. Calcium folinate 400mg/m2 intravenous infusion (over 2 hours or more), on the first day, followed by 5-fluorouracil 400mg/m2 intravenous bolus injection, then continuous intravenous infusion of 1200mg/m2/day for 2 days.
  Arms: SC0191 + 5-FU/LV

SUMMARY:
The goal of this clinical trial is to evaluate the preliminary safety and efficacy of SC0191 as single agent or in combination with bevacizumab or 5-FU/LV in advanced colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily participate in the clinical study and sign an informed consent form;
2. Male or female subjects aged ≥18 years;
3. Subjects diagnosed with stage IV colorectal cancer confirmed by histology or cytology and not suitable for curative surgical treatment;
4. Subjects who have previously received fluoropyrimidine-based chemotherapy, oxaliplatin, and irinotecan with or without anti-EGFR or anti-VEGF targeted therapy, and experienced disease progression or intolerance to the most recent treatment regimen; the number of prior lines of systemic antitumor therapy for advanced colorectal cancer does not exceed 2 lines;
5. ECOG performance status of 0 to 1;
6. Expected survival of ≥3 months;
7. At least one measurable lesion according to RECIST 1.1 criteria, defined as a lesion with a longest diameter ≥10 mm on CT scan or MRI (excluding lymph nodes) or a short diameter ≥15 mm for lymph nodes. Lesions located in previously irradiated or otherwise locally treated areas are generally not considered measurable unless there is documented disease progression;
8. Adequate organ function and bone marrow hematopoietic function;
9. Fertile subjects (both male and female) must agree to use a reliable method of contraception (hormonal or barrier method, or abstinence) with their partners for at least 6 months from the time of signing the informed consent form until the last dose of the study drug; female subjects of childbearing potential must have a negative pregnancy test within 14 days before the first use of the investigational drug.

Exclusion Criteria:

1. Subjects known to be MSI-H who have not received immunotherapy;
2. Subjects with spinal cord compression, symptomatic/unstable brain metastases, or leptomeningeal metastases. Exclusion: Subjects with stable symptoms of brain metastases after prior treatment (completion of definitive radiotherapy and/or surgery, cessation of corticosteroid therapy, and stable symptoms for at least 14 days);
3. Subjects with radiological evidence of tumor invasion or encasement of major vessels (Cohort A);
4. Subjects with uncontrollable pleural effusion, ascites, or pericardial effusion at screening;
5. Subjects with a history of other malignant tumors within 5 years prior to study drug initiation, except for early-stage tumors cured by curative treatment, such as basal cell carcinoma or squamous cell carcinoma of the skin, cervical carcinoma in situ, ductal carcinoma in situ of the breast, superficial bladder cancer, localized prostate cancer, etc.;
6. Subjects with significant cardiovascular diseases, including NYHA class II-IV heart failure, congestive heart failure, second-degree or higher atrioventricular block, myocardial infarction within the past 6 months, unstable arrhythmias or angina, significant QT interval prolongation (baseline-corrected QTc interval >470 milliseconds on ECG), stroke within the past 6 months, or PTCA (percutaneous transluminal coronary angioplasty) or CABG (coronary artery bypass grafting) within the past 6 months;
7. Subjects with poorly controlled hypertension;
8. Subjects with viral infectious diseases at screening meeting the following criteria:
9. HIV seropositivity;
10. Hepatitis B: HBsAg positivity with HBV-DNA quantification above the upper limit of normal;
11. Hepatitis C: HCV antibody positivity with HCV-RNA quantification above the upper limit of normal;
12. Subjects with active infections requiring systemic antimicrobial therapy as judged by the investigator, deemed unsuitable for participation in this study;
13. Subjects who have undergone allogeneic tissue/organ transplantation;
14. Subjects with malabsorption syndrome or other gastrointestinal abnormalities that may significantly affect oral drug absorption (such as ulcerative lesions, uncontrollable nausea, vomiting, diarrhea, malabsorption syndrome, and small bowel resection, etc.);
15. Subjects with hereditary bleeding or coagulation disorders, or a history of severe non-traumatic bleeding, or a history of ineffective platelet transfusion (within the past 1 year before initial study drug administration), or any disease that significantly increases the risk of bleeding;
16. Subjects with a history of any of the following during treatment with Bevacizumab-based regimens (or biosimilars): venous or arterial thromboembolic events, gastrointestinal perforation, grade 4 hypertension, grade 3 proteinuria, or grade 3 or higher bleeding events (Cohort A).
17. Subjects who have undergone major surgery, open biopsy, or experienced severe traumatic injury within 28 days before first use of the investigational drug, or are expected to undergo major surgery during the study. Subjects who have undergone minor surgery within 7 days before first use of the investigational drug, such as fine needle aspiration or core biopsy. Subjects with a history of esophageal varices or bleeding peptic ulcer within 3 months before first use of the investigational drug (Cohort A).
18. Known history of dihydropyrimidine dehydrogenase (DPD) deficiency. History of discontinuing fluoropyrimidine treatment due to ≥3 grade diarrhea (Cohort B).
19. Subjects with a history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis requiring corticosteroid treatment, or any clinical evidence suggesting active interstitial lung disease;
20. Subjects diagnosed with autoimmune diseases during screening or receiving long-term systemic corticosteroid therapy (dose exceeding 10 mg/day of prednisone or equivalent) or any other form of immunosuppressive therapy due to autoimmune diseases;
21. Subjects whose toxicity from prior anticancer therapy has not resolved to ≤ grade 1 (CTCAE 5.0) (excluding alopecia, decreased hearing, and stable endocrine disorders treated with alternative therapies);
22. Subjects previously treated with WEE1 inhibitors;
23. Subjects with a history of hypersensitivity reactions to SC0191, Bevacizumab (Cohort A), fluoropyrimidines (Cohort B), calcium folinate (Cohort B) active ingredients, or their inactive excipients or similar drugs;
24. Subjects who received radiation therapy to more than 25% of the bone marrow area within 28 days before first use of the investigational drug;
25. Subjects vaccinated with live vaccines within 28 days before first use of the investigational drug.
26. Subjects who received chemotherapy, biologic therapy, endocrine therapy, or other antitumor therapy within 28 days before first use of the investigational drug; or received small molecule targeted therapy within 28 days or 5 half-lives (whichever is shorter) before first use of the investigational drug; or received traditional Chinese medicine for antitumor therapy within 7 days before first use of the investigational drug;
27. Subjects who received systemic corticosteroids (prednisone equivalent >10 mg/day) or other immunosuppressive therapy within 14 days before first use of the investigational drug, except for local, ocular, intra-articular, intranasal, and inhalational corticosteroid therapy; or received corticosteroids for prophylactic treatment (e.g., prevention of contrast agent allergy) ;
28. Subjects who received moderate or potent inhibitors of CYP3A4 (such as amprenavir, atazanavir, boceprevir, clarithromycin, conivaptan, darunavir, diltiazem, erythromycin, foscarnet, indinavir, itraconazole, ketoconazole, lopinavir, mibefradil, miconazole, nefazodone, nelfinavir, posaconazole, ritonavir, telithromycin, verapamil, voriconazole, etc.) or moderate or potent inducers of CYP3A4 (such as carbamazepine, felbamate, nevirapine, phenobarbital, phenytoin, primidone, rifampin, efavirenz, modafinil, etc.) within 14 days before first use of the investigational drug;
29. Subjects who require regular use of proton pump inhibitors (PPIs) during the study or received PPI therapy within 14 days before first use of the investigational drug (such as omeprazole, esomeprazole, lansoprazole, pantoprazole, and rabeprazole, etc.);
30. Subjects who require long-term therapeutic doses of anticoagulants or antiplatelet drugs (prophylactic use of low-dose anticoagulants is allowed, provided that the anticoagulation parameters specified in the inclusion criteria are met); low-dose anticoagulants may be used to maintain venous catheter patency;
31. Subjects with psychiatric disorders or poor compliance;
32. Pregnant or lactating female subjects;
33. Subjects whom the investigator considers to have other serious systemic medical history, or for other reasons are not suitable for participation in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 12 months
Incidence and Severity of Dose Limiting Toxicities (DLTs) | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No